CLINICAL TRIAL: NCT04042467
Title: Greenlight Plus Study: A Randomized Study of Approaches to Early Childhood Obesity Prevention
Brief Title: Greenlight Plus Study: Approaches to Early Childhood Obesity Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Duke University (Other); University of North Carolina, Chapel Hill (Other); Stanford University (Other); NYU Langone Health (Other); University of Miami (Other); Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Bill Heerman, Assistant Professor, Internal Medicine and Pediatrics, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 190311
Record Dates: First submitted 2019-07-19; First posted 2019-08-02 (Actual); Results first posted 2025-10-16 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-09

CONDITIONS: Behavior, Health; Child Obesity
MeSH Terms: conditions — Health Behavior; Pediatric Obesity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: All Greenlight Plus personnel that are in a position to change the study protocol or its implementation in study participants should be blinded to information that may allow them to do so, from when the study starts until the study ends, with specific exceptions. This means that all investigators and study staff should be blinded to study data aggregated by study arm that have the potential to impact the study's outcome.
  The study statistician and programmers s/he designates will be unblinded to post-randomization outcome, mediator, moderator and process data for the purposes of generating DSMB reports.
  The study statistician will remain objective when carrying out the activities of conducting the trials - preparing randomization schemes, processing of the data, cleaning and editing the data, preparation of analyses/reports of outcome, mediator, moderator and blinded process data, and transmitting those data to the DSMB.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Greenlight Plus (Experimental): Families will receive the Greenlight intervention plus a health information technology (HIT) intervention aimed at supporting family goal-setting and behavior change.
  This design allows us to determine if HIT and the asynchronous support it provides between well-child visits can promote additional behavior change and obesity prevention.
  Interventions: Behavioral: Greenlight Plus; Behavioral: Greenlight
- Greenlight (Active Comparator): During each of the recommended well child visits from 0-24 months, pediatric residents, trained in clear health communication skills and shared goal-setting, will use the Greenlight Toolkit of low literacy, age- specific, parent education booklets to promote healthy family behaviors and obesity prevention.
  Interventions: Behavioral: Greenlight

INTERVENTIONS:
Behavioral: Greenlight Plus — Families randomized to the Greenlight Plus arm will receive a HIT intervention starting at the newborn clinic visit. During the newborn visit, these families will receive basic instructions on how to access the Greenlight technology platform, which includes the iOTA text-messaging application and a website (usable on desktop or mobile platform). Families will receive text messages and goal-setting over the first 2 years of the child's life.
  Arms: Greenlight Plus
Behavioral: Greenlight — All residents and families seen in the participating clinics will receive the basic Greenlight materials.

SUMMARY:
A randomized controlled trial enrolling 900 parent-infant dyads (English and Spanish speaking) comparing Greenlight (control), a behavioral intervention focusing on nutrition, physical activity, media use, and sleep as compared to Greenlight Plus (intervention) which includes the above materials plus a health information technology (HIT) intervention aimed at supporting family goal-setting and behavior change during well-child checks throughout the first 2 years of life.

DETAILED DESCRIPTION:
The investigators propose a randomized trial to compare the effectiveness of two different approaches to early childhood obesity prevention in children 0-2 years of age. The investigators will randomize 900 parent-infant dyads, recruited from six newborn nurseries/primary care clinics. The participating organizations are part of both CORNET, a national practice-based research network of pediatric residency primary care practices supported by the Academic Pediatric Association (APA), and PCORnet, the national research network supported by PCORI. In the nursery or at the first newborn clinic visit, eligible families will be consented and randomized to one of two arms. In Arm 1 ("Greenlight"), during each of the recommended well child visits from 0-24 months, pediatric residents, trained in clear health communication skills and shared goal-setting, will use the Greenlight Toolkit of low literacy, age-specific, parent education booklets to promote healthy family behaviors and obesity prevention. In Arm 2 ("Greenlight Plus"), families will receive the Greenlight intervention plus a health information technology (HIT) intervention aimed at supporting family goal-setting and behavior change. This design allows us to determine if HIT and the asynchronous support it provides between well-child visits can promote additional behavior change and obesity prevention.

Specific Aims & Hypotheses (H) include:

Aim 1: Compare the effectiveness of the 2 arms on weight-for-length and other weight measures through age 2.

H1: Arm 2 will be significantly better than Arm 1 in supporting healthy child weight-for-length trajectory over 2 years;

Aim 2: Compare the effectiveness of the two approaches on parent-reported outcomes, including child feeding and physical activity behaviors, parent feeding beliefs and behaviors, media use, and quality of doctor-patient communication.

H2: Arm 2 will be significantly better at improving parent-reported health behaviors.

Aim 3: Examine differences in main outcomes by social determinants, including race/ethnicity, language, health literacy.

H3: A literacy- and culturally-sensitive approach to obesity prevention will result in equal subgroup improvements.

Aim 4: To compare weight-for-length trajectory over 2 years in both intervention arms with a non-enrolled comparison group, using data from the PCORnet Common Data Model at participating sites.

H4: PCORnet analysis will reveal the benefit of both Greenlight approaches (Arms 1 and 2) compared to before Greenlight intervention implementation and the added benefit of Arm 2 (Greenlight Plus) over other approaches.

ELIGIBILITY:
Inclusion Criteria:

For this study, eligible caregiver/infant dyads will be those with:

1. an English- or Spanish-speaking parent/legal guardian,
2. infant born in the newborn nursery with plans to have care in the local clinic OR presenting in that clinic for the first newborn visit (1-21 days of life),
3. attendance at first newborn clinic visit
4. no plans to leave the clinic within 2 years
5. Completion of baseline data collection (survey data, child weight and length measures prior to randomization).
6. Own a smartphone with access to data services

Exclusion Criteria:

Infant exclusion criteria:

1. born prior to 34 weeks gestation or birth weight <1500 grams; weight <3rd %tile at enrollment (World Health Organization growth curves); or
2. any chronic medical problem that may affect weight gain (e.g., metabolic disease, uncorrected congenital heart disease, renal disease, high-calorie formula; cleft palate; Down syndrome).

Caregiver exclusion criteria include:

1. <18 years old;
2. serious mental or neurologic illness that impairs ability to consent/participate;
3. poor visual acuity (corrected vision worse than 20/50 with Rosenbaum Screener).
4. biological mother is HIV-positive

Max Age: 21 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 900 (Actual)
Dates: Start 2019-11-06 (Actual); Primary Completion 2024-01-17 (Actual); Study Completion 2024-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Russell Rothman, MD, MPP, Principal Investigator — Vanderbilt University Medical Center; William Heerman, MD, MPH, Principal Investigator — Vanderbilt University Medical Center; Charles Wood, MD, MPH, Principal Investigator — Duke University; Kori Flower, MD, MS, MPH, Principal Investigator — University of North Carolina, Chapel Hill; Lee Sanders, MD, MPH, Principal Investigator — Stanford University; H. Shonna Yin, MD, MS, Principal Investigator — NYU School of Medicine, NYU Langone Health; Alan Delamater, PhD, Principal Investigator — University of Miami; Eliana Perrin, MD, MPH, Principal Investigator — Johns Hopkins University
Locations (6):
- United States (6):
  - Stanford University, Stanford, California
  - University of Miami, Coral Gables, Florida
  - New York University, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee

REFERENCES:
- [Background] Heerman WJ, Perrin EM, Yin HS, Schildcrout JS, Delamater AM, Flower KB, Sanders L, Wood C, Kay MC, Adams LE, Rothman RL. The Greenlight Plus Trial: Comparative effectiveness of a health information technology intervention vs. health communication intervention in primary care offices to prevent childhood obesity. Contemp Clin Trials. 2022 Dec;123:106987. doi: 10.1016/j.cct.2022.106987. Epub 2022 Oct 30. PMID 36323344
- [Result] Heerman WJ, Rothman RL, Sanders LM, Schildcrout JS, Flower KB, Delamater AM, Kay MC, Wood CT, Gross RS, Bian A, Adams LE, Sommer EC, Yin HS, Perrin EM; Greenlight Investigators; de la Barrera B, Bility M, Cruz Jimenez Smith M, Cruzatte EF, Guevara G, Howard JB, Lampkin J, Orr CJ, Pilotos McBride J, Quintana Forster L, Ramirez KS, Rodriguez J, Schilling S, Shepard WE, Soto A, Velazquez JJ, Wallace S. A Digital Health Behavior Intervention to Prevent Childhood Obesity: The Greenlight Plus Randomized Clinical Trial. JAMA. 2024 Dec 24;332(24):2068-2080. doi: 10.1001/jama.2024.22362. PMID 39489149

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from medical clinics at six medical centers: Duke University, University of Miami, New York University Grossman School of Medicine/Bellevue Hospital Center, University of North Carolina at Chapel Hill, Stanford University, and Vanderbilt University Medical Center. Study enrollment occurred between November 2019 and August 2021.
Pre-assignment Details: Enrollment numbers and number of participants Started/Completed represent the number of dyads (child and parent).
Period: Overall Study
Arm/Group | Greenlight Plus | Greenlight
Started (The numbers reported in the table represent dyads (child and parent). The number of individual participants in the Greenlight Plus group was n=898 (449 children and 449 parents), and the number of individual participants in the Greenlight group was n=902 (451 children and 451 parents).) | 449 | 451
Completed (The numbers reported in the table represent dyads (child and parent). The number of individual participants who completed the study in the Greenlight Plus group was n=770 (385 children and 385 parents), and the number of individual participants who completed the study in the Greenlight group was n=784 (392 children and 392 parents)) | 385 | 392
Not Completed | 64 | 59

BASELINE CHARACTERISTICS:
Population: The number of individual participants in the Greenlight Plus group was n=898 (449 children and 449 parents), and the number of individual participants in the Greenlight group was n=902 (451 children and 451 parents).
Groups:
- Total: Total of all reporting groups
Arm/Group | Greenlight Plus | Greenlight | Total
Number analyzed (Participants) | 898 | 902 | 1800
Age, Customized [Median (Inter-Quartile Range); unit: weeks] — Child gestational age (weeks) Population: Data is for the gestational age of children only. Data missing for 1 Greenlight Plus participant.
  weeks
    Child gestational age: number analyzed (Participants) | 448 | 451 | 899
    Child gestational age | 39.3 [38.6 to 40.0] | 39.1 [38.4 to 40.0] | 39.1 [38.4 to 40.0]
Age, Customized [Median (Inter-Quartile Range); unit: years] — Population: Data is for the age of parents only.
  years
    Parent age: number analyzed (Participants) | 449 | 451 | 900
    Parent age | 30.2 [25.6 to 34.2] | 30.1 [25.6 to 34.4] | 30.1 [25.6 to 34.3]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex of child-Female | 243 | 233 | 476
  Sex of child-Male | 206 | 218 | 424
  Sex of parent-Female | 433 | 441 | 874
  Sex of parent-Male | 15 | 10 | 25
  Sex of parent-Other | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Data missing for 2 Greenlight Plus participants.
  Participants
    Child race/ethnicity: number analyzed (Participants) | 447 | 451 | 898
    Child race/ethnicity: Black, non-Hispanic | 62 | 81 | 143
    Child race/ethnicity: Hispanic | 204 | 201 | 405
    Child race/ethnicity: White, non-Hispanic | 95 | 90 | 185
    Child race/ethnicity: Other or multiple | 86 | 79 | 165
    Parent race/ethnicity: number analyzed (Participants) | 449 | 451 | 900
    Parent race/ethnicity: Black, non-Hispanic | 68 | 85 | 153
    Parent race/ethnicity: Hispanic | 230 | 215 | 445
    Parent race/ethnicity: White, non-Hispanic | 104 | 100 | 204
    Parent race/ethnicity: Other or multiple | 47 | 51 | 98
Child birth weight [Median (Inter-Quartile Range); unit: kg] — Population: Data missing for 1 Greenlight Plus participant.
  kg
    number analyzed (Participants) | 448 | 451 | 899
    (all) | 3.3 [3.1 to 3.6] | 3.3 [3.0 to 3.6] | 3.3 [3.0 to 3.6]
Parent health literacy [Count of Participants; unit: Participants] — Parent health literacy was assessed by the Newest Vital Sign 6-item literacy screening tool. A score greater than or equal to 4 was categorized as adequate. Population: Data missing for 13 Greenlight Plus and 16 Greenlight participants.
  Participants
    number analyzed (Participants) | 436 | 435 | 871
    Adequate | 186 | 185 | 371
    Limited | 250 | 250 | 500
Parent preferred language [Count of Participants; unit: Participants] — Population: Data is for the preferred language of parents only
  Participants
    number analyzed (Participants) | 449 | 451 | 900
    Spanish | 155 | 158 | 313
    English | 294 | 293 | 587
Parent education level [Count of Participants; unit: Participants] — Population: Data is for the education level of parents only
  Participants
    number analyzed (Participants) | 449 | 451 | 900
    No school | 1 | 2 | 3
    Grade school (K-4) | 5 | 4 | 9
    Middle school (5-8) | 26 | 39 | 65
    Some high school (9-12) | 58 | 60 | 118
    High school graduate or GED | 127 | 101 | 228
    Some college or technical/vocational school | 76 | 81 | 157
    College degree | 90 | 100 | 190
    Post graduate or professional degree | 66 | 64 | 130
Annual household income [Count of Participants; unit: Participants] — Population: Data is for the income of the household
  Participants
    number analyzed (Participants) | 449 | 451 | 900
    <$20,000 | 114 | 103 | 217
    $20,000 to $49,000 | 115 | 108 | 223
    $50,000 to $99,999 | 42 | 58 | 100
    $100,000 or more | 64 | 60 | 124
    Do not know/not sure | 91 | 96 | 187
    Prefer not to answer | 23 | 26 | 49
Household food insecurity [Count of Participants; unit: Participants] — Food insecurity was assessed by the 6-item US Department of Agriculture measure. A score greater than or equal to 2 was categorized as food insecure. Population: Data is for the household. Data missing from 3 Greenlight Plus and 3 Greenlight households.
  Participants
    number analyzed (Participants) | 446 | 448 | 894
    Food insecure | 67 | 74 | 141
    Food secure | 379 | 374 | 753

OUTCOME MEASURES:

1. Primary Outcome: Child Weight for Length Trajectory
Description: The primary outcome was child weight for length (kg/m) trajectory over 2 years. Weight and length measurements were obtained during pediatric care visits and abstracted from the medical record.
Time Frame: Baseline to 24 months
Population: Follow-up outcome measures were not obtained for 3 Greenlight Plus participants and 1 Greenlight participant.
  NOTE: While the analysis included data from children (n=896) and their parents (n=896), the unit of analysis was the child. Therefore, the number of participants has been reported consistently across the Participant Flow, Baseline Characteristics, and Outcome Measures sections.
Measure: Mean (Standard Deviation); unit: kg/m
Arm/Group | Greenlight Plus | Greenlight
Number analyzed (Participants) | 446 | 450
kg/m
  1 Month: number analyzed (Participants) | 259 | 271
  1 Month | 8.0 (0.9) | 8.0 (0.8)
  2 Months: number analyzed (Participants) | 410 | 405
  2 Months | 9.3 (1.0) | 9.4 (1.0)
  4 Months: number analyzed (Participants) | 380 | 375
  4 Months | 10.8 (1.2) | 11.0 (1.2)
  6 Months: number analyzed (Participants) | 372 | 378
  6 Months | 11.9 (1.2) | 12.0 (1.3)
  9 Months: number analyzed (Participants) | 355 | 364
  9 Months | 12.7 (1.3) | 12.9 (1.3)
  12 Months: number analyzed (Participants) | 346 | 337
  12 Months | 13.1 (1.3) | 13.4 (1.5)
  15 Months: number analyzed (Participants) | 294 | 319
  15 Months | 13.5 (1.4) | 13.8 (1.6)
  18 Months: number analyzed (Participants) | 323 | 349
  18 Months | 13.9 (1.4) | 14.2 (1.6)
  24 Months: number analyzed (Participants) | 380 | 387
  24 Months | 14.8 (1.6) | 15.2 (2.0)
Statistical Analysis 1: Comparison: Greenlight Plus vs Greenlight; Linear mixed-effects model (random intercepts and slopes for clinics and participants within clinics). A priori adjustment for baseline variables: child birth weight and biological sex, race/ethnicity, health literacy, language, education, income, and food insecurity. Child age and birth weight were included using natural splines with 3 DoF. Effect evaluated using Wald test with a 2-sided, 0.05 significance level. Null hypothesis: Equal weight-for-length growth trajectories in the two groups; Test type: Superiority; p < 0.001, Regression, Linear — The p-value was not adjusted for multiple comparisons, and the a priori threshold for statistical significance was 0.05; Wald test (4 DoF) of intervention main effect and 3 intervention by age interaction parameters equal 0 vs. alternative that at least one was not 0; Estimated intervention effect at 24 mo. = -0.33, 95% CI 2-sided [-0.57 to -0.09] — The p-value is for the Wald test (4 DoF) evaluating whether the Greenlight Plus and Greenlight group trajectories were significantly different. The estimation parameter is the model-estimated intervention effect at 24 months (kg/m)

2. Secondary Outcome: Child BMI Z-score Trajectory
Time Frame: Baseline to 24 months
Reporting Status: Not Posted

3. Secondary Outcome: Child Weight-for-length Z-score Trajectory
Time Frame: Baseline to 24 months
Reporting Status: Not Posted

4. Secondary Outcome: Child Overweight and/or Obesity
Description: Outcome defined by CDC or WHO standards
Time Frame: at 24 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data were collected across the study's 2-year duration for each participant.
Description: AE: Any unfavorable and unintended sign, symptom, laboratory abnormality, or disease associated with study participation.
  SAE: Is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in death or persistent or significant disability/incapacity, or is a congenital anomaly/birth defect in the offspring of a participant.
  A study-related event follows a temporal sequence from participation and cannot be reasonably explained by other factors.
Arm/Group | Greenlight Plus | Greenlight
All-Cause Mortality (participants affected / at risk) | 0/898 | 2/902
Serious Adverse Events (participants affected / at risk) | 0/898 | 0/902
Other Adverse Events (participants affected / at risk) | 1/898 | 0/902
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Greenlight Plus (N=898) | Greenlight (N=902)
(General disorders) | 1 | 0 — Participant selected "yes" to an AE in a self-administered survey. Study team unable to reach participant for further info. Believed to be a misclick but unable to confirm. Case accepted by IRB with no requested changes to protocol.

LIMITATIONS AND CAVEATS:
Some population groups were underrepresented or not represented (e.g., patients who did not prefer to speak English or Spanish). The study was unable to collect reliable data on web-based dashboard use, limiting the ability to evaluate which digital components of the Greenlight Plus intervention were associated with effectiveness. Anthropometric measures collected during clinical care may be susceptible to measurement error. However, annual training was implemented to minimize errors.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-04): https://cdn.clinicaltrials.gov/large-docs/67/NCT04042467/Prot_SAP_000.pdf